CLINICAL TRIAL: NCT00110747
Title: A Randomized, Double-Blind, Placebo Controlled, Paired Study Evaluating the Efficacy of S-Caine™ Peel (Lidocaine 7% and Tetracaine 7% Cream) in Providing Local Dermal Anesthesia for Non-Ablative Facial Laser Resurfacing in Adults
Brief Title: S-Caine™ Peel (Skin Numbing Cream) to Treat Pain During Non-Ablative Facial Laser Resurfacing in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ZARS Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCP-41-05
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- S-Caine Peel (Experimental)
  Interventions: Drug: S-Caine™ Peel (lidocaine and tetracaine topical cream 7%/7%)
- Placebo Peel (Placebo Comparator)
  Interventions: Drug: Placebo Peel

INTERVENTIONS:
Drug: S-Caine™ Peel (lidocaine and tetracaine topical cream 7%/7%) — S-Caine Peel comprising a 1:1 eutectic mixture of 7% lidocaine and 7% tetracaine was applied topically. A thin layer of the peel (approximately 1 mm in thickness) was applied and remained on the treatment area for 30 minutes (±2 minutes).
  Other Names: Pliaglis
  Arms: S-Caine Peel
Drug: Placebo Peel — Peel was applied topically. A thin layer of the peel (approximately 1 mm in thickness) was applied and remained on the treatment area for 30 minutes (±2 minutes).
  Other Names: Placebo
  Arms: Placebo Peel

SUMMARY:
Lasers are used for non-ablative resurfacing of facial rhytides, atrophic scars, and a variety of epidermal and dermal lesions. Pain associated with the non-ablative laser treatment has been described as moderate to severe. For this reason, local anesthesia is commonly used to eliminate or minimize the pain. S-Caine™ Peel (lidocaine 7% and tetracaine 7% cream) is a eutectic formulation of lidocaine and tetracaine. The purpose of this study is to evaluate if S-Caine Peel is effective in providing topical local dermal anesthesia for non-ablative facial laser resurfacing in adults.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, placebo-controlled, paired study that evaluated the effectiveness of S-Caine Peel in providing local dermal anesthesia for non-ablative facial laser resurfacing. Patients received a concurrent application of S Caine Peel and placebo for 30 minutes (±2 minutes).

Patients who presented to the study site for a non-ablative facial laser resurfacing and who met study entry criteria were invited to participate in the study. At the screening visit, the study, including potential risks and benefits, was clearly explained to each patient, and written informed consent was obtained. A medical history was obtained including skin type, demographic data, prior and current medical disorders, and the use of concomitant medications. A brief physical examination was performed including taking basic vital signs and examining the skin at the study drug application site. If applicable, a urine pregnancy test was performed. The screening visit could occur on the same day as the procedure visit.

At the procedure visit, patients were randomized to receive a 30-minute (±2 minute) application of S Caine Peel either on the right or left treatment area and to receive a concurrent 30-minute (±2 minutes) application of placebo on the alternate treatment area. The point of reference was always the patient's right and left. S-Caine Peel and placebo were dispensed to cover the treatment area with a uniform thickness of approximately 1 mm. Study drug was applied to the right treatment area first, then concurrently to the left treatment area. Similarly, the study drug was removed first from the right treatment area and then from the left treatment area. Following removal of the study drugs, the investigator or physician subinvestigator evaluated each study drug application site for erythema, edema, blanching or other skin reactions. The right treatment area was evaluated first, followed by the left treatment area.

After the skin evaluations, the laser procedure was performed on the right treatment area, followed by patient and investigator efficacy evaluations for the right treatment area. The laser procedure was then performed on the left treatment area, followed by patient and investigator efficacy evaluations for the left treatment area.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years of age or older
* Patient elects to undergo non-ablative facial laser resurfacing procedure

Exclusion Criteria:

* Patient is pregnant or breastfeeding
* Patient has participated in a clinical trial of an unapproved drug within the previous 30 days
* Patient has participated in any previous clinical trial involving S-Caine Peel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Patient's evaluation of pain | 30 minutes
  Patient's evaluation of pain using a 100 mm Visual Analog scale (VAS)

SECONDARY OUTCOMES:
Number of participants with adverse events | 30 minutes
  To monitor the nature and frequency of adverse events (AEs) associated with the application of S-Caine Peel

CONTACTS AND LOCATIONS:
Overall Officials: Tina Alster, MD, Principal Investigator — Washington Institute of Dermatologic Laser Surgery
Locations (3):
- United States (3):
  - Midwest Cutaneous Research, Clinton Township, Michigan
  - Laser and Skin Surgery Center of New York, New York, New York
  - New York Dermatology, New York, New York